CLINICAL TRIAL: NCT02843438
Title: Evaluation of Biological Biomarkers Diagnostic of Toxoplasmosis Uveitis
Acronym: BIOLUVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 38RC09.014
Record Dates: First submitted 2016-07-21; First posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Subjects Clinically Suspected an Active Source of Toxoplasmosis Chorioretinitis Infection
Keywords: Toxoplasmosis; Uveitis; Chorioretinitis; Infection
MeSH Terms: conditions — Toxoplasmosis; Uveitis; Chorioretinitis; Infections | interventions — Punctures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects suspected of toxoplasmosis chorioretinitis infection (Other): Subjects clinically suspected at least of one active source of toxoplasmosis chorioretinitis infection
  Interventions: Other: Fluorescein angiography; Other: Dilated fundus examination; Biological: Toxoplasmosis serology; Drug: Anti-toxoplasmosis treatment; Drug: Anti-inflammatory treatments; Other: Puncture in anterior chamber

INTERVENTIONS:
Other: Fluorescein angiography
Other: Dilated fundus examination
Biological: Toxoplasmosis serology
Drug: Anti-toxoplasmosis treatment
Drug: Anti-inflammatory treatments
Other: Puncture in anterior chamber

SUMMARY:
Toxoplasmosis affects one to two newborn each 10000 births. Among them, 1 to 2 % develop learning disabilities or die, and 4 to 27 % develop a chorioretinitis sometimes leading to an amblyopia responsible for visual impairment. Toxoplasmosis uveitis affects too adults immunocompetent and immunodepressed who have had an acquired toxoplasmosis. Clinical diagnosis of ocular toxoplasmosis is more complicated in presence of posterior neuro-retinitis, inflammation of the papilla, uveitis without chorioretinitis, fuchs heterochromic iridocyclitis, scleritis, diffuse necrotizing or multifocal retinitis. In this situation biological markers diagnostic and prognostic of toxoplasmosis uveitis are useful.

Highly kept molecules (during evolution) like stress proteins (Hsp) are are found in the host and the pathogen and there can trigger a crossed immune response. Stress proteins haven't been explored yet, in the context of toxoplasmosis uveitis on humans.

The hypothesis is that Hsp70 and antibodies anti-Hsp70 are diagnostic and prognostic markers of ocular toxoplasmosis.

The goal is to evaluate diagnosis value of biological markers (Hsp70 and antibodies IgG anti-Hsp70) in toxoplasmosis uveitis.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Subjects clinically suspected at least of one active source of toxoplasmosis chorioretinitis infection
* Persons affiliated to national social security

Exclusion Criteria:

* Pregnant, parturient or breastfeeding women
* Persons deprived of liberty by judicial or administrative decision, person under legal protection
* Refusal by a patient to do the PCA (anterior chamber puncture)
* Patients whose following will be difficult or nonexistent

Max Age: 18 Years | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2010-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
ELISA tests | About an hour
  ELISA (enzyme linked immunosorbent assay) tests. Biological markers evaluation : stress protein Hsp70 and antibodies anti-Hsp70.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Bouillet, Professor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Bonfioli AA, Orefice F. Toxoplasmosis. Semin Ophthalmol. 2005 Jul-Sep;20(3):129-41. doi: 10.1080/08820530500231961. PMID 16282146
- [Background] Bouillet L, Sarrot-Reynauld F, Gonzalvez B, Massot C, Romanet J, Mouillon M. [Diagnostic strategy in uveitis: a prospective study in 125 cases]. J Fr Ophtalmol. 2000 Jun;23(6):569-75. French. PMID 10880922
- [Background] Brenier-Pinchart MP, Morand-Bui V, Fricker-Hidalgo H, Equy V, Marlu R, Pelloux H. Adapting a conventional PCR assay for Toxoplasma gondii detection to real-time quantitative PCR including a competitive internal control. Parasite. 2007 Jun;14(2):149-54. doi: 10.1051/parasite/2007142149. PMID 17645187
- [Background] Chen M, Aosai F, Norose K, Mun HS, Yano A. The role of anti-HSP70 autoantibody-forming V(H)1-J(H)1 B-1 cells in Toxoplasma gondii-infected mice. Int Immunol. 2003 Jan;15(1):39-47. doi: 10.1093/intimm/dxg004. PMID 12502724
- [Background] Chumpitazi BF, Boussaid A, Pelloux H, Racinet C, Bost M, Goullier-Fleuret A. Diagnosis of congenital toxoplasmosis by immunoblotting and relationship with other methods. J Clin Microbiol. 1995 Jun;33(6):1479-85. doi: 10.1128/jcm.33.6.1479-1485.1995. PMID 7650171
- [Background] Chumpitazi BF, Bouillet L, Drouet MT, Kuhn L, Garin J, Zarski JP, Drouet C. Biological autoimmunity screening in hepatitis C patients by anti-HepG2 lysate and anti-heat shock protein 70.1 autoantibodies. Eur J Clin Microbiol Infect Dis. 2009 Feb;28(2):137-46. doi: 10.1007/s10096-008-0599-y. Epub 2008 Aug 12. PMID 18696130
- [Background] Delair E, Monnet D, Grabar S, Dupouy-Camet J, Yera H, Brezin AP. Respective roles of acquired and congenital infections in presumed ocular toxoplasmosis. Am J Ophthalmol. 2008 Dec;146(6):851-5. doi: 10.1016/j.ajo.2008.06.027. Epub 2008 Aug 23. PMID 18723143
- [Background] Derouin F, Bultel C, Roze S. (Coordination rédactionnelle). Toxoplasmose: état des connaissances et évaluation du risque lié à l'alimentation. Rapport du groupe de travail " Toxoplasma gondii " de l'Afssa. Coordination éditoriale : Thomann C & Ribeiro F. AFSSA Déc. 2005, pp318.
- [Background] Desmonts G. Definitive serological diagnosis of ocular toxoplasmosis. Arch Ophthalmol. 1966 Dec;76(6):839-51. doi: 10.1001/archopht.1966.03850010841012. No abstract available. PMID 5924940
- [Background] Direskeneli H, Saruhan-Direskeneli G. The role of heat shock proteins in Behcet's disease. Clin Exp Rheumatol. 2003 Jul-Aug;21(4 Suppl 30):S44-8. PMID 14727460
- [Background] Echeverria PC, Matrajt M, Harb OS, Zappia MP, Costas MA, Roos DS, Dubremetz JF, Angel SO. Toxoplasma gondii Hsp90 is a potential drug target whose expression and subcellular localization are developmentally regulated. J Mol Biol. 2005 Jul 22;350(4):723-34. doi: 10.1016/j.jmb.2005.05.031. PMID 15967463
- [Background] Fang H, Aosai F, Mun HS, Norose K, Ahmed AK, Furuya M, Yano A. Anaphylactic reaction induced by Toxoplasma gondii-derived heat shock protein 70. Int Immunol. 2006 Oct;18(10):1487-97. doi: 10.1093/intimm/dxl081. Epub 2006 Aug 30. PMID 16943259
- [Background] Holland GN. Reconsidering the pathogenesis of ocular toxoplasmosis. Am J Ophthalmol. 1999 Oct;128(4):502-5. doi: 10.1016/s0002-9394(99)00263-9. PMID 10577593
- [Background] Imamura Y, Kurokawa MS, Yoshikawa H, Nara K, Takada E, Masuda C, Tsukikawa S, Ozaki S, Matsuda T, Suzuki N. Involvement of Th1 cells and heat shock protein 60 in the pathogenesis of intestinal Behcet's disease. Clin Exp Immunol. 2005 Feb;139(2):371-8. doi: 10.1111/j.1365-2249.2005.02695.x. PMID 15654837
- [Background] Kodjikian L, Wallon M, Fleury J, Denis P, Binquet C, Peyron F, Garweg JG. Ocular manifestations in congenital toxoplasmosis. Graefes Arch Clin Exp Ophthalmol. 2006 Jan;244(1):14-21. doi: 10.1007/s00417-005-1164-3. Epub 2005 May 20. PMID 15906073
- [Background] Lyons RE, Johnson AM. Heat shock proteins of Toxoplasma gondii. Parasite Immunol. 1995 Jul;17(7):353-9. doi: 10.1111/j.1365-3024.1995.tb00902.x. PMID 8552407
- [Background] Maubon D, Ajzenberg D, Brenier-Pinchart MP, Darde ML, Pelloux H. What are the respective host and parasite contributions to toxoplasmosis? Trends Parasitol. 2008 Jul;24(7):299-303. doi: 10.1016/j.pt.2008.03.012. Epub 2008 May 29. PMID 18514029
- [Background] Pelloux H, Mouillon M, Romanet JP, Reynier P, Ligeon P, Goullier-Fleuret A, Ambroise-Thomas P. [Ocular toxoplasmosis. Comparison between two biological methods to study aqueous humor]. Presse Med. 1991 Oct 26;20(34):1655-8. French. PMID 1836568
- [Background] Quintana FJ, Cohen IR. Heat shock proteins as endogenous adjuvants in sterile and septic inflammation. J Immunol. 2005 Sep 1;175(5):2777-82. doi: 10.4049/jimmunol.175.5.2777. PMID 16116161
- [Background] SenGupta D, Norris PJ, Suscovich TJ, Hassan-Zahraee M, Moffett HF, Trocha A, Draenert R, Goulder PJ, Binder RJ, Levey DL, Walker BD, Srivastava PK, Brander C. Heat shock protein-mediated cross-presentation of exogenous HIV antigen on HLA class I and class II. J Immunol. 2004 Aug 1;173(3):1987-93. doi: 10.4049/jimmunol.173.3.1987. PMID 15265933
- [Background] Silva NM, Gazzinelli RT, Silva DA, Ferro EA, Kasper LH, Mineo JR. Expression of Toxoplasma gondii-specific heat shock protein 70 during In vivo conversion of bradyzoites to tachyzoites. Infect Immun. 1998 Aug;66(8):3959-63. doi: 10.1128/IAI.66.8.3959-3963.1998. PMID 9673286
- [Background] Wang XH, Qin Y, Hu MH, Xie Y. Dendritic cells pulsed with gp96-peptide complexes derived from human hepatocellular carcinoma (HCC) induce specific cytotoxic T lymphocytes. Cancer Immunol Immunother. 2005 Oct;54(10):971-80. doi: 10.1007/s00262-005-0662-9. Epub 2005 Jun 18. PMID 15965645